CLINICAL TRIAL: NCT04256096
Title: Randomization of Endovascular Treatment With Stent-retriever and/or Thromboaspiration vs. Best Medical Therapy in Acute Ischemic Stroke Due to Large VEssel OcclusioN Trial in the Extended Time Window
Brief Title: Randomization of Endovascular Treatment in Acute Ischemic Stroke in the Extended Time Window
Acronym: RESILIENTExt
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Hospital das Clínicas de Ribeirão Preto (Other); Hospital Geral de Fortaleza (Other Government); Hospital de Base (Other); Federal University of São Paulo (Other); Fundação Faculdade Regional de Medicina de São José do Rio Preto (Other); UPECLIN HC FM Botucatu Unesp (Other); University of Campinas, Brazil (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); Universidade Federal do Paraná (Other); Hospital Estadual Central (Unknown); Hospital Sao Jose do Avai (Unknown); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Federal University of Uberlandia (Other); Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Responsible Party: Principal Investigator, SHEILA CRISTINA OURIQUES MARTINS, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17877519.6.1001.5327
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Ischemic
Keywords: stroke; ischemic stroke; thrombectomy; treatment; acute stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: The randomization employs a 1:1 ratio of mechanical thrombectomy with stent-retriever and/or thromboaspiration versus medical management alone
Who Masked: Outcomes Assessor
Masking Description: Sham endovascular procedure has been rejected due to the medical risk of the angiography and practical issues that difficult to maintain blindness of investigators. For the primary endpoint, subjects will be followed for 90 days post-randomization. Distribution of the modified Rankin Scale scores at 90 days will be evaluated by two separate assessors who are blinded to treatment. Primary Endpoint will consider central core lab readings only (video interview with RFA method) with local reading as a back-up mechanism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thrombectomy (Experimental): mechanical thrombectomy with stent-retriever and/or thromboaspiration
  Interventions: Device: Thrombectomy
- Clinical treatment (Active Comparator): Best Medical treatment
  Interventions: Device: Thrombectomy

INTERVENTIONS:
Device: Thrombectomy — Endovascular treatment of large vessel occlusion (mechanical thrombectomy) with stent-retriever and/or thromboaspiration (neurointerventionalist choice)
  Other Names: Endovascular treatment

SUMMARY:
A phase III, randomized, multi-center, open label clinical trial that will examine whether endovascular treatment is superior to standard medical therapy alone in patients who suffer a large vessel anterior circulation ischemic stroke within 8-24 hours from time last seen well

DETAILED DESCRIPTION:
Prospective, multi-center, randomized, controlled, open-label, blinded-endpoint trial with a sequential design. The randomization employs a 1:1 ratio of mechanical thrombectomy with stent-retriever and/or thromboaspiration versus medical management alone in patients who suffer a large vessel anterior circulation ischemic stroke between 8 and 24 hours from time last seen well. Randomization will be done under a minimization process using age (≤68 vs. >68 years), baseline NIHSS (<17 v. ≥17), ASPECTS (5-7 vs. 8-10), therapeutic window (6-12 or 12-24 hours after TLKW), occlusion site (Intracranial ICA or M1), and clinical site. For the primary endpoint, subjects will be followed for 90 days post-randomization. Sham endovascular procedure has been rejected due to the medical risk of the angiography and practical issues that difficult to maintain blindness of investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke where patient is ineligible for IV thrombolytic treatment or the treatment is contraindicated (e.g., subject presents beyond recommended time from symptom onset), or where patient has received IV thrombolytic therapy without clinical improvement.
2. No significant pre-stroke functional disability (mRS ≤2)
3. Baseline NIHSS score obtained prior to randomization must be equal or higher than 8 points (assessed within one hour prior to qualifying imaging)
4. Age ≥18 years (no upper age limit)
5. Occlusion (TICI 0-1) of the intracranial ICA (distal ICA or T occlusions) and/or MCA-M1 segment suitable for endovascular treatment, as evidenced by CTA, MRA or angiogram, with or without concomitant cervical carotid occlusion or stenosis.
6. The presence of Age-Adjusted modified Clinical ASPECTS Mismatch (mCAM) defined as ASPECTS 5-10 and one of the following criteria:

   1. NIHSS ≥ 8 and >50% involvement in 0-1 Cortical (e.g. M1-6) ASPECTS areas (any age);
   2. NIHSS ≥ 8 and >50% involvement in 0-2 Cortical (e.g. M1-6) ASPECTS areas (and age < 80 years old);
   3. NIHSS ≥ 15 and >50% involvement in 0-3 Cortical (e.g. M1-6) ASPECTS areas (and age < 80 years old).
7. Patient treatable within 6-24 hours of symptom onset. Symptoms onset is defined as point in time the patient was last seen well (at baseline). Treatment start is defined as arterial puncture.
8. Informed consent obtained from patient or acceptable patient surrogate

Exclusion Criteria:

-Clinical criteria

1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
2. Baseline platelet count < 30.000/µL
3. Baseline blood glucose of < 50mg/dL
4. Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using AHA guidelines recommended medication (including iv antihypertensive drips), the patient can be enrolled.
5. Patients in coma defined as totally unresponsive; responding only with reflexes or being areflexic (Intubated patients for transfer could be randomized only in case an NIHSS is obtained by a neurologist prior transportation).
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS
7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
8. History of life-threatening allergy (more than rash) to contrast medium
9. Subjects who has received IV t-PA treatment beyond 4.5 hours from the beginning of the symptoms
10. Woman of childbearing potential who is known to be pregnant or who has a positive pregnancy test on admission.
11. Subject participating in a study involving an investigational drug or device that would impact this study.
12. Cerebral vasculitis
13. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤2. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
14. Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).

    - Neuroimaging criteria
15. Hypodensity on CT or restricted diffusion on MRI amounting to an ASPECTS score of <5.
16. Complete involvement of more than 3 cortical ASPECTS areas (e.g. M1, M2, M3, M4, M5, or M6).
17. Complete absence of leptomeningeal collaterals on CT angiography (e.g. Malignant CTA pattern or score 0).
18. CT or MR evidence of hemorrhage (the presence of GRE microbleeds is allowed).
19. Significant mass effect with midline shift.
20. Evidence of ipsilateral carotid occlusion, high grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment
21. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation)
22. Evidence of intracranial tumor (except small meningioma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale scores | 90 days
  Distribution of the modified Rankin Scale scores at 90 days (shift analysis). The score range from zero to 6 with higher values indicating a worst functional outcome at 90 days

SECONDARY OUTCOMES:
Proportion of Patients with Functional independence in 90 days | 90 days
  Functional independence defined as mRS ≤2
Disability on the utility-weighted modified Rankin scale (UW-mRS) | 90 days
  Mean score for disability on the utility-weighted modified Rankin scale (UW-mRS). The score range from 1 to zero with higher values indicating a better functional outcome at 90 days
Quality of life measured by EuroQol Group 5-Dimension Self-Report Questionnaire (EuroQol / EQ5D) | 90 days and 1 year
  Quality of life analysis as measured by EuroQol/EQ5D 5-Dimension Self-Report Questionnaire, on which scores range from -0.176 to 1, with higher values indicating a better quality of life]) at 90 days
Mortality at 90 days | 90 days
  Mortality at 90 days
Proportion of patients with Intracranial Hemorrhage at 24 hours | 24 hours
  Clinically significant ICH rates at 24 (-2/+12) hours. All intracerebral hemorrhages will be classified by a central core-lab using the Heidelberg criteria. Symptomatic ICH will be defined as per the SITS-MOST definition: deterioration in NIHSS score of ≥4 points within 24 hours from treatment and evidence of intraparenchymal hemorrhage type 2 in the 22 to 36 hours follow-up imaging scans.
Procedural related complications | immediately after procedure
  Procedural related complications: arterial perforation, arterial dissection, and embolization in a previously uninvolved vascular territory

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — Emory University; Sheila CO Martins, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (14):
- Brazil (14):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Associacao Congregacao de Santa Catarina, Vitória, Espírito Santo
  - Hospital de Base, Brasília, Federal District
  - Hospital das Clínicas de Uberlândia, Uberlândia, Minas Gerais
  - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Conferencia Sao jose do Avai, Itaperuna, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre - ISCMPA, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Hospital de Clínicas - UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas de Ribeirao Preto, Ribeirão Preto, São Paulo
  - Fundacao Faculdade Regional de Medicina S J Rio Preto, São José do Rio Preto, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual de Sao Paulo, São Paulo, São Paulo
  - Universidade Federal de São Paulo - UNIFESP/EPM, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Because of the sensitive nature of the data collected for this study, requests to access the dataset from qualified researchers trained in human subject confidentiality protocols may be sent to the principal investigators
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after de publication for 6 months
Access Criteria: Because of the sensitive nature of the data collected for this study, requests to access the dataset from qualified researchers trained in human subject confidentiality protocols may be sent to the principal investigators

REFERENCES:
- [Derived] Roaldsen MB, Lindekleiv H, Mathiesen EB. Intravenous thrombolytic treatment and endovascular thrombectomy for ischaemic wake-up stroke. Cochrane Database Syst Rev. 2021 Dec 1;12(12):CD010995. doi: 10.1002/14651858.CD010995.pub3. PMID 34850380